CLINICAL TRIAL: NCT07145008
Title: Suprachoroidal Triamcinolone in Macular Edema for Patients With Non-Infectious Uveitis Resistant to Subtenon Triamcinolon
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Mutar, Medical Doctor, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-234
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Macular Edema (ME); Non Infectious Uveitis
Keywords: Suprachoroidal Triamcinolone; Macular Edema; Non infectious uveitis; Subtenon resistant
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Suprachoroidal Triamcinolone treatment arm (Experimental)
  Interventions: Drug: Suprachoroidal triamcinolone acetonide injection

INTERVENTIONS:
Drug: Suprachoroidal triamcinolone acetonide injection — For suprachoroidal injection, we developed a custom-made delivery system to access the potential suprachoroidal space. A 1 mL tuberculin syringe fitted with a 27-gauge needle was prepared, and a plastic sleeve from a 24-26 G IV cannula was placed over the needle as a spacer to control penetration depth.

SUMMARY:
The goal of this study is to learn if a suprachoroidal triamcinolone injection can treat vision-threatening swelling in the center of the retina (macular edema) caused by non-infectious uveitis, especially in people who did not improve after a standard steroid injection around the eye (sub-Tenon injection).

The main questions it aims to answer are:

Does vision improve on the eye chart after the injection?

Does the injection lower retinal swelling (reduction in thickness) within 3 months?

Participants will:

Have a pre-treatment check (vision test, slit-lamp exam, and a retinal scan called OCT).

Receive one suprachoroidal triamcinolone injection under anesthetics drops in a sterile setting (operating room) with standard monitoring.

Return for visits about 1 month and 3 months after treatment for repeat vision tests, and OCT scans.

Contact the clinic if they notice pain, redness, new floaters, or worsening vision.

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious uveitis complicated with macular edema
* Uveitic macular edema of less than four months' duration
* Macular edema persisted despite lack of intra-ocular inflammation
* No response to posterior sub-Tenon triamcinolone acetonide injections

Exclusion Criteria:

* Those with epiretinal membrane-associated macular edema
* Below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity improvement | 3 months
  visual acuity improvement was defined as a gain of two or more lines in visual acuity or a reduction in logMAR values

SECONDARY OUTCOMES:
Central Macular Thickness | 3 Months
  A reduction in central macular thickness (CMT) exceeding 20%.

CONTACTS AND LOCATIONS:
Locations (1):
- Ibn Al-Haitham Eye Teaching Hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT07145008/Prot_SAP_000.pdf